CLINICAL TRIAL: NCT00599534
Title: A Randomized Double Blind Controlled Trial on the Effect of Treatment in Children With Obstructive Sleep Apnea Syndrome.
Brief Title: Controlled Trial on Effect of Montelukast Treatment in Children With Obstructive Sleep Apnea Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator has transferred to another Institution
Sponsor: University of Louisville (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB# 07.0135
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 4 mg tablet for 16 weeks
  Interventions: Drug: Montelukast
- 2 (Placebo Comparator): 5 mg for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — 4 mg oral tablets
  Arms: 1
Drug: Placebo — 5mg tablets
  Arms: 2

SUMMARY:
Oral therapy with montelukast may lead to improved polysomnographic findings in children with mild to moderate OSAS with and without allergic rhinitis who a priori require T&A for OSAS.

- A significant proportion of the children with OSAS treated with montelukast will show reduced severity of OSAS, and this will obviate the need for surgical T&A.

DETAILED DESCRIPTION:
Primary Specific Aim. To conduct a randomized double blind 16-week trial comparing the effect on polysomnographic measures of the administration of once a day oral montelukast therapy vs. placebo in children with OSAS.

Secondary Specific Aim. For all children with the original AHI at diagnosis of >2 hrTST, we expect improvements in the severity of sleep apnea to occur following treatment with montelukast. Therefore, we will examine the overall reduction in AHI and also how many of these children have AHI< 2 after the 16-week treatment. In other words, the percentage of children converting from needing T&A surgery before treatment with montelukast to not needing surgery after treatment will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic snoring children > 2 years of age and < 10 years of age, who snore and have an apnea hypopnea index (AHI) >2/hrTST (hour total sleep time), and in whom T&A is therefore contemplated. Also among these, we will include children referred for evaluation for snoring who have a history of allergic rhinitis.

Exclusion Criteria:

* Hypersensitivity to montelukast
* Immunodeficiency or immunosuppressant therapy
* Craniofacial, neuromuscular, syndromic or defined genetic abnormalities
* Acute upper respiratory tract infection
* Systemic corticosteroid therapy or antibiotic therapy in the 2 weeks previous to the study
* Children who already had adenotonsillectomy.

In addition, children chronically receiving oral antihistamine preparations or nasal decongestants will be required to continue using these medications throughout the duration of the study. Patients receiving immunotherapy will continue on the same regimen without escalation of dose and frequency throughout the duration of the study. In addition, patients with severe OSA who in the opinion of their treating physicians require early surgical intervention for their OSA will be excluded from eligibility to the study.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of children converting from needing T&A surgery before treatment with montelukast to not needing surgery after treatment will be examined. | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: Leila Kheirandish, M.D., Principal Investigator — University of Louisville; Lelia Kheirandish, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - University of Louisville Pediatric Sleep Medicine Center, Louisville, Kentucky
  - University of Louisville Pediatrics Sleep Medicine Center, Louisville, Kentucky

REFERENCES:
- [Derived] Kheirandish-Gozal L, Bandla HP, Gozal D. Montelukast for Children with Obstructive Sleep Apnea: Results of a Double-Blind, Randomized, Placebo-Controlled Trial. Ann Am Thorac Soc. 2016 Oct;13(10):1736-1741. doi: 10.1513/AnnalsATS.201606-432OC. PMID 27439031